CLINICAL TRIAL: NCT02706431
Title: Evaluation of Oxygenation by 100% Oxygen Via High Flow Nasal Cannula During Apnea in Adult Elective Surgical ENT Patients
Brief Title: Oxygenation by 100% Oxygen Via High Flow Nasal Cannula in Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Jonsson Fagerlund, Associate Professor/Senior Consultant, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Apnoic Oxygenation
Record Dates: First submitted 2015-12-15; First posted 2016-03-11 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Anaesthesia, General; Anesthesia, Intravenous; Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normoventilation (No Intervention): The patients will be normoventilated before anesthesia
- Hyperventilation (Experimental): Prior to anesthesia, the patients will hyperventilate during 2 mins or until symptoms from the central nervous system (e.g. dizziness).
  Interventions: Procedure: Hyperventilation

INTERVENTIONS:
Procedure: Hyperventilation
  Arms: Hyperventilation

SUMMARY:
Oxygenation with high-flow nasal cannula with 100% oxygen has only been evaluated in a limited number of studies. Although data are convincing it is of importance to evaluate this new concept in our department before implementing it into clinical practice.

The general purpose of this project is to evaluate a new ventilation strategy during ENT-surgery based on oxygenation with high-flow nasal cannula with 100% oxygen with focus on gas exchange.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, >18 years old
2. ENT-surgery where apnea is of benefit for the surgeon (eg. intraoral or laryngeal surgery) and the anesthesia time is <40 mins.
3. Capable of understanding the study information and sign the written consent.

Exclusion Criteria:

1. ASA>2
2. NYHA >2
3. BMI >30
4. Pregnancy
5. Manifest cardiac failure or coronary disease
6. Neuromuscular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Change in arterial carbon dioxide (pCO2) | From start of anaesthesia to end of apnoea oxygenation or max 30 minutes
Change in arterial pH | From start of anaesthesia to end of apnoea oxygenation or max 30 minutes
Change in arterial oxygen tension (pO2) | From start of anaesthesia to end of apnoea oxygenation or max 30 minutes

SECONDARY OUTCOMES:
Does hyperventilation prior to anaesthesia and apnoea oxygenation cause any difference in pCO2 in the end of the apnea (i.e. at up to 30 minutes) compared to normoventilation? | In the end of the apnoea period, i.e. at approximately 20 minutes
Does hyperventilation prior to anaesthesia and apnoea oxygenation cause any difference in pH in the end of the apnea (i.e. at up to 30 minutes) compared to normoventilation? | In the end of the apnoea period, i.e. at approximately 20 minutes
Does hyperventilation prior to anaesthesia and apnoea oxygenation cause any difference in pO2 in the end of the apnea (i.e. at up to 30 minutes) compared to normoventilation? | In the end of the apnoea period, i.e. at approximately 20 minutes
Does the high oxygen content cause atelectasis measures as change in relation between pCO2 and end tidal carbon dioxide | Until discharge from the postoperative unit, often max 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, MD, PhD, Principal Investigator — Karolinska University Hospital and Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gustafsson IM, Lodenius A, Tunelli J, Ullman J, Jonsson Fagerlund M. Apnoeic oxygenation in adults under general anaesthesia using Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) - a physiological study. Br J Anaesth. 2017 Apr 1;118(4):610-617. doi: 10.1093/bja/aex036. PMID 28403407